CLINICAL TRIAL: NCT07029178
Title: A Randomized Controlled Trial on Taurine's Therapeutic Effect on Acute Radiation-induced Oral Mucositis and Dermatitis
Brief Title: Taurine's Therapeutic Effect on Acute Radiation-induced Oral Mucositis and Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Yue He, MD, Section head, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JYKQ-2025-001
Record Dates: First submitted 2025-05-21; First posted 2025-06-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Radiation Induced Oral Mucositis; Radiodermatitis
Keywords: double-blind; randomized controlled trial; taurine; radiodermatitis; radiation-induced oral mucositis
MeSH Terms: conditions — Radiodermatitis | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Doctors, patients and clinical research coordinator (CRC) are blind. The medicine will be encoded before the beginning of the trial, and will be administered before each radiotherapy session by CRC. After the patient take the medication, the CRC takes the patient to the treatment room for radiotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): From the first day of radiotherapy to the end of radiotherapy, the control group was treated with 24 grams of placebo before each day's radiotherapy.
  Interventions: Drug: Placebo granule
- Taurine group (Experimental): From the first day of radiotherapy to the end of radiotherapy, the experimental group was treated with 24 grams of taurine granule (containing 4.8 grams of taurine) before each day's radiotherapy.
  Interventions: Drug: Taurine granule

INTERVENTIONS:
Drug: Taurine granule — 24 grams of taurine granule + 2 Gray radiation dose each time.
  Other Names: Radiotherapy
  Arms: Taurine group
Drug: Placebo granule — 24 grams of placebo granule + 2 Gray radiation dose each time.
  Other Names: Radiotherapy
  Arms: Control group

SUMMARY:
This is a single-center, double-blind, randomized controlled study. The patients were divided into control group and experimental group, 80 cases each. From the first day of radiotherapy to the end of radiotherapy, the experimental group was treated with 24 grams of taurine granule (containing 4.8 grams of taurine) before each day's radiotherapy. The control group was treated with the same amount of placebo.

DETAILED DESCRIPTION:
Implementation of double-blind:

Doctors, patients and clinical research coordinator (CRC) are blind. The medicine will be encoded before the beginning of the trial, and will be administered before each radiotherapy session by CRC. After the patient take the medication, the CRC takes the patient to the treatment room for radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily joined the study, were informed of the purpose and process of the study, signed the informed consent form, and were willing and able to abide by the study protocol.
2. Aged 18 to 80, with no gender restrictions.
3. Patients that require radiotherapy after surgery for oral/oropharyngeal cancer. After evaluation by the radiation oncologist, radiotherapy at 30 sessions /60Gy is planned.
4. The expected survival period is more than 6 months.
5. No radiotherapy for the head and neck has been performed in the past, and no other medications that affect the results of this trial have been used. No chemotherapy or immunotherapy was performed within one month before the beginning of the trial.

Exclusion criteria:

1. Uncontrollable local or systemic infections of the oral cavity and head and neck.
2. Active or history of autoimmune diseases; Diseases requiring systemic steroid hormones or immunosuppressive medications.
3. Bleeding occurred within 3 months before enrollment, including but not limited to: gastrointestinal bleeding caused by gastric fundus or esophageal varices, increased risk of bleeding caused by portal hypertension, active gastrointestinal bleeding, etc. Or there is a risk of major bleeding as assessed by the researcher.
4. Arterial/venous thrombosis that occurred within 6 months prior to the screening, such as cerebrovascular accidents, deep vein thrombosis and pulmonary embolism, etc.
5. Interstitial pneumonia or active pneumonia with clinical significance, or other respiratory diseases that seriously affect lung function.
6. History of cardiovascular diseases, including but not limited to: (1) Congestive heart failure (NYHA grade > 2); (2) Unstable angina pectoris; (3) Myocardial infarction occurred in the past three months; (4) Any supraventricular arrhythmia or ventricular arrhythmia that requires treatment or intervention.
7. Severe endocrine or hematopoietic system diseases (such as diabetes, leukemia, etc.), gastrointestinal obstruction, active bleeding, gastric perforation and other conditions.
8. Combined with malignant tumors of other organs.
9. Intractable or refractory epilepsy, with a large amount of pleural effusion, ascites, pericardial effusion, etc. that cannot be controlled by medicines.
10. History of HIV, syphilis, active hepatitis, active pulmonary tuberculosis, active EBV and/or CMV infection within one year before screening, or those with a history of active pulmonary tuberculosis infection for more than one year without regular treatment; active hepatitis B or C. Patients with positive HBsAg or HBcAb can participate in this study if the HBV DNA test is below the lower limit of the normal value detected by the research center; patients with positive HCV antibody can participate in this study if the HCV RNA test is below the lower limit of the normal value detected by the research center.
11. History of allogeneic bone marrow transplantation or solid organ transplantation.
12. Have received cell therapy products that have undergone genetic modification or editing in the past.
13. Have previously used medicines that can cause medication-related osteonecrosis of the jaw.
14. Have taken drugs containing taurine within one month before randomization in this study.
15. Allergic to taurine.
16. Patients who, in addition to radiotherapy, requires chemotherapy or immunotherapy simultaneously.
17. Mental illness, alcohol abuser, drug user or drug abuser.
18. Pregnant or lactating women; Women who plans to become pregnant within half a year after treatment.
19. Poor compliance or other circumstances assessed by the researcher as unsuitable for participation in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate and severity of acute radiation-induced oral mucositis | Day 0 (before the first radiotherapy),7,14,21,28,35,42 (after the last radiotherapy),49±1 (follow-up),56±2 (follow-up),70±5 (follow-up), 126±5 (study endpoint).
  The severity of acute radiation-induced oral mucositis is evaluated by RTOG (Radiation Therapy Oncology Group) classification. The subjective feeling of radiation-induced oral mucositis is evaluated via the weekly oral mucositis questionnaire during radiotherapy.

SECONDARY OUTCOMES:
Incidence rate and severity of acute radiodermatitis | Day 0 (before the first radiotherapy),7,14,21,28,35,42 (after the last radiotherapy),49±1 (follow-up),56±2 (follow-up),70±5 (follow-up), 126±5 (study endpoint).
  The severity of acute radiodermatitis is evaluated by RTOG (Radiation Therapy Oncology Group) classification.
Number of participants with Safety physiological parameters | Clinical symptoms and adverse events are recorded when occured. Blood routine and blood biochemistry examination are evaluated during screening and on day 14, 28, 42 and 70±5d.
  The safety of placebo granule and taurine granule is evaluated by clinical symptoms, adverse events (assessed by CTCAE v5.0), blood routine examination (including red blood cells, hemoglobin, blood platelet, white blood cell, basophilic granulocyte, Eosinophils, lymphocyte, mononuclear leucocyte, neutrophil, c reactive protein, procalcitonin, etc.), blood biochemistry examination (including alanine transaminase, glutamic-pyruvic transaminase, alkaline phosphatase, total protein, albumin, total bilirubin, direct bilirubin, blood urea nitrogen, creatinine, potassium ion, sodion, chloridion, calcium ion, magnesium ion, etc.), etc.

OTHER OUTCOMES:
Immunological parameters of peripheral blood | The blood immunoglobulin and CD molecule examination will be conducted during screening, on day 42 (the end of radiotherapy) and on day 70±5d.
  The immunomodulatory effects of placebo granule and taurine granule is evaluated by blood immunoglobulin examination (IgA、IgG、IgE、IgM) and blood CD molecule (CD3、CD4、CD8、CD16、CD19、CD56) examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China